CLINICAL TRIAL: NCT05661526
Title: The Effect of Game-Based Activity on Knowledge and Persistence in Blood Transfusion in Nursing Students: A Randomized Controlled Trial
Brief Title: The Effect of Game-Based Activity on Blood Transfusion in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Lutfiye Nur Uzun, PhD Student, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AIBU-HEM-UZUN-002
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: Blood Transfusion; Nursing Education; Board Game

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled study with experimental and control groups consisting of pre-test, post-test and persistence test.
Who Masked: Outcomes Assessor
Masking Description: Outcome evaluations will be conducted by a researcher blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bloodpoly board game (Experimental): Students in the Bloodpoly board game group; In the designated classroom and common time frame and under the supervision of researchers, they will be provided with an average of 50 minutes of board games per day for three days. For this, four groups of five students will be formed and students will be randomly assigned to these groups. Students will then be asked to move on to the four areas where the board game takes place. Four groups will start playing Bloodpoly simultaneously. The game will continue until all questions are finished.
  Interventions: Other: Bloodpoly board game
- Text-to-speech group (Active Comparator): Students in the text-to-speech group; 50 minutes of reading time will be organized per day for three days in the designated classroom and common time and under the supervision of the researchers During the reading time, the content of the topic related to blood transfusion described by the researchers will be given to the students and they will be provided with reading. At the end of the period, the documents given will be taken back by the researchers.
  Interventions: Other: Text-to-speech group

INTERVENTIONS:
Other: Bloodpoly board game — Blood transfusion training given by Bloodpoly board game
  Arms: Bloodpoly board game
Other: Text-to-speech group — Blood transfusion training given by text-to-speech
  Arms: Text-to-speech group

SUMMARY:
The aim of this randomized controlled study, which included pre-test, posttest and perseverance test, was to determine the effect of game-based learning on nursing students' knowledge levels about blood transfusion, to determine the permanence level of learning and satisfaction with the training method.

The fundamental question it aims to answer is:

•Does the blood transfusion training given to nursing students by the board game playing method have an effect on the level of knowledge, the permanence of the information and satisfaction with the training method? Participants will participate in an educational activity related to blood transfusion. The researchers will compare whether the blood transfusion training given to nursing students with the board game playing method is effective or not with the text-reading method.

DETAILED DESCRIPTION:
Students who meet the criteria for inclusion in the study and agree to participate in the study will be divided into experimental and control groups using the computer-aided randomization system. After randomization, the appropriate time frame will be determined by taking into account the course schedules with the students. During the common time frame, students will be informed about the research and asked to fill out the Informed Consent Forms. The subject of blood transfusion (KGI: 1.00), which was prepared by the researchers and sent to five academic nurses who are experts in the field for scope validity, will be transferred to the students in three course hours (150 minutes) in the form of theoretical training and power point presentation. Within the scope of theoretical training, students; the structure of blood and blood, the functions of blood, the combination of blood, blood groups, Rh factor, blood products, blood transfusion, blood transfusion indications, safe blood transfusion, basic points in the transfusion process of blood and blood products, blood transfusion process steps and blood transfusion reactions will be explained. After the lecture is completed, "Blood Transfusion Information Test" and Personal Information Form will be applied to the students.

After the theoretical part of the course is completed, the application part is carried out differently for the control and experimental group and after the application of the control group is finished, the application of the experimental group will be carried out.

Students in the control group; 50 minutes of reading time will be organized per day for three days in the designated classroom and common time and under the supervision of the researchers During the reading time, the content of the topic related to blood transfusion described by the researchers will be given to the students and they will be provided with reading. At the end of the period, the documents given will be taken back by the researchers. This practice will continue for three days and at the end of the third day, "Blood Transfusion Knowledge Test" and "Satisfaction with Educational Methods" will be applied to the students.

The students in the experimental group; In the designated classroom and common time frame and under the supervision of researchers, they will be provided with an average of 50 minutes of board games per day for three days. For this, four groups of five students will be formed and students will be randomly assigned to these groups. Students will then be asked to move on to the four areas where the board game takes place. Four groups will start playing Bloodpoly simultaneously. The game will continue until all questions are finished. After the Bloodpoly game, "Blood Transfusion Knowledge Test" and "Satisfaction Survey from Educational Methods" will be applied to the students.

Three weeks after the application of the Control and Experimental group is completed, the "Blood Transfusion Knowledge Test" will be re-administered to all students to measure persistence in the level of knowledge.

Board Game The board game called Bloodpoly was inspired by the game Monopoly when it was designed. Bloodpoly is a board game for nursing students with information questions about blood transfusion. The game is built on a square cardboard floor. The questions and "surprise" contents in the "one-on-one", "short short", "true-false", "what am I?", "attention!" sections in the blood transfusion information test were written on cards prepared in different colors. Surprise card contents include commands such as "ask your opponent a question", "go back to the beginning", "donate a blood", which add excitement to the game. The player who comes to the black "Bankruptcy" box on the game track must donate all the blood in his hand to the blood center. The cards are randomly placed in the middle of the track, above their own color. The Bloodpoly game consists of a total of 70 boxes. The boxes are painted in 10 "one-on-one" green, 10 "short short" pink, 10 "right-wrong" purple, 10 "what am I?" blue, 10 "attention!" red, 10 "surprise" yellow, and 10 "bankruptcy" black. Colors are randomly placed on the track. There is a "start" box representing the start of the track. In the middle of the track there is a blood bank where players can buy blood products. In the blood bank there are cards in the form of blood bags representing the blood product. There are icons of different characters in the game to represent the players and to see their progress on the track. Advancements in the game are made by throwing a single dice consisting of six numbers.

ELIGIBILITY:
Inclusion Criteria:

* To be a second year student of the nursing department
* To be eligible to participate in the curriculum research
* Not having received any previous training in blood transfusions
* Not having clinical experience in the subject
* Volunteering to participate in the study

Exclusion Criteria:

* Not being eligible to participate in curriculum research
* Have any previous training in blood transfusion
* Have clinical experience in the subject
* Not volunteering to participate in the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Nursing students' knowledge of blood transfusion: First test | Just before application
  "Blood Transfusion Knowledge Test" is a test prepared by researchers by scanning the literature and includes 50 questions of blood transfusion. The test consists of five sections and each section contains 10 questions. The total score, which is calculated by summing the scores obtained from the five sections of the test, constitutes the participant's blood transfusion knowledge level score. The total score that can be reached in the test varies between 0-75.

SECONDARY OUTCOMES:
Nursing students' knowledge of blood transfusion: Second test | Immediately after application
  "Blood Transfusion Knowledge Test" is a test prepared by researchers by scanning the literature and includes 50 questions of blood transfusion. The test consists of five sections and each section contains 10 questions. The total score, which is calculated by summing the scores obtained from the five sections of the test, constitutes the participant's blood transfusion knowledge level score. The total score that can be reached in the test varies between 0-75.
Satisfaction levels of nursing students with the training method | Immediately after application
  "Satisfaction with Educational Methods Survey" "Satisfaction with Educational Methods Survey" is a questionnaire developed by Gürpınar and consists of 16 propositions (Cronbach alpha: 0.84). Each proposition is scored on a scale of 1 to 5 according to the 5-point lique. In the survey, at least 16 and at most 80 points are given to the satisfaction of the students from the educational methods It is determined that the satisfaction levels of the students increase as the score obtained from the survey increases, and the satisfaction levels decrease as they decrease

OTHER OUTCOMES:
Nursing students' knowledge of blood transfusion: Persistence test | Three weeks after application
  "Blood Transfusion Knowledge Test" is a test prepared by researchers by scanning the literature and includes 50 questions of blood transfusion. The test consists of five sections and each section contains 10 questions. The total score, which is calculated by summing the scores obtained from the five sections of the test, constitutes the participant's blood transfusion knowledge level score. The total score that can be reached in the test varies between 0-75.

CONTACTS AND LOCATIONS:
Overall Officials: Lütfiye Nur Uzun, PhD Student, Principal Investigator — Bolu Abant İzzet Baysal University Faculty of Health Sciences Nursing Department; Birgül Cerit, Assoc.Prof., Principal Investigator — Bolu Abant İzzet Baysal University Faculty of Health Sciences Nursing Department
Locations (1):
- Bolu Abant İzzet Baysal University Faculty of Health Sciences Nursing Department, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.